CLINICAL TRIAL: NCT02277210
Title: Effect of Follicular Flushing on the Ongoing Pregnancy Rate in Patients Who Developed Four or Fewer Follicles of 14mm Following Standard Ovarian Stimulation for In-vitro Fertilization Treatment - A Randomized Controlled Trial.
Brief Title: Follicular Flushing in Patients With Suboptimal Responses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ernest Hung-Yu Ng, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW14-428
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — flushing solution PBSuc 50

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-flushing group (Placebo Comparator): Aspiration alone for all follicular larger than 10mm on both sides. Follicular fluid and flushing will be examined by the embryologists to identify any oocytes.
  Interventions: Other: Flushing
- Flushing group (Active Comparator): aspiration of follicles that are larger than 10 mm on both sides followed by follicular flushing for up to 4 times. Follicular fluid and flushing will be examined by the embryologists to identify any oocytes.
  Interventions: Other: Flushing

INTERVENTIONS:
Other: Flushing — aspiration of follicles that are larger than 10 mm on both sides followed by follicular flushing for up to 4 times. Follicular fluid and flushing will be examined by the embryologists to identify any oocytes.

SUMMARY:
The aim of the present study is to determine the effect of follicular flushing on the ongoing pregnancy rate in patients who developed four or fewer follicles of 14mm following standard ovarian stimulation for IVF.

DETAILED DESCRIPTION:
Oocyte aspiration under the guidance of transvaginal ultrasound is an integral part in IVF treatment. Follicular flushing has been advocated. However, subsequent data from randomized trials failed to demonstrate any benefits with routine follicular flushing in normally responding patients. Instead, it has been shown to prolong the operating time, increase the procedure-related pain and analgesics requirement. Most of the IVF centers no longer perform routine follicular flushing in normally responding patients.

The potential role of follicular flushing in patients with a limited number of developing follicles is conflicting based on the recently published randomized trials. The aim of the present study is to determine the effect of follicular flushing on the ongoing pregnancy rate in patients who developed four or fewer follicles of 14mm following standard ovarian stimulation for IVF.

ELIGIBILITY:
Inclusion Criteria:

1. Age of women <43 years
2. Normal uterine cavity on saline sonogram
3. Endometrial thickness >=8mm on the day of hCG

Exclusion Criteria:

1. Planned not to have fresh embryo transfer
2. Cycle cancelled prior to hCG administration
3. Natural cycle IVF
4. Presence of hydrosalpinges on scanning which are not surgically treated
5. Presence of endometrial polyps on scanning
6. Undergoing preimplantation genetic diagnosis

Max Age: 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-06-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 10 weeks of gestation

SECONDARY OUTCOMES:
number of oocytes retrieved | on the day of retrieval
number of embryo available for transfer | on the day of embryo transfer
clinical pregnancy rate | 6 weeks of gestation
operation time of the retrieval | on the day of retrieval
pain score of retrieval | on the day of retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ernest Ng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Georgiou EX, Melo P, Cheong YC, Granne IE. Follicular flushing during oocyte retrieval in assisted reproductive techniques. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD004634. doi: 10.1002/14651858.CD004634.pub4. PMID 36409927